CLINICAL TRIAL: NCT06190041
Title: Kinesiophobia in Patients With Chronic Low Back Pain: an Evaluation on Relevant Factors and Its Effects on Quality of Life
Brief Title: Kinesiophobia in Patients With Chronic Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Duygu Karamanlıoğlu, Principal investigator, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMEAH-KAEK 2023/37
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Kinesiophobia; Disability; Quality of Life
Keywords: chronic low back pain; Kinesiophobia; Disability
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Low back pain is an important health problem that is common in public and causes serious socio-economic losses. Low back pain that persists for more than 12 weeks is defined as chronic low back pain. The prognosis in patients with chronic low back pain is generally not good and it significantly affects the patient's daily living activities and workforce. In the clinical course of chronic low back pain, patients generally reduce some activities or avoid them altogether due to fear of pain or concern about worsening of the initial lesion. This fear is called "kinesiophobia", which is an important factor in the chronicity of low back pain and the resulting functional disabilities. Kinesiophobia causes loss of flexibility, decreased muscle performance, muscle wasting, and all of these lead to a decrease in social and physical activities, which perpetuates and aggravates the disability. The aim of this study is to determine the relationship between the frequency of kinesiophobia in chronic low back pain patients and age, gender, body mass index, educational status, occupation, pain intensity and disability, and to examine the effect of kinesiophobia on quality of life.

DETAILED DESCRIPTION:
Approximately 200 patients with chronic low back pain lasting ≥12 weeks between the ages of 18-75 who applied to the outpatient clinic will be included in the study. Demographic data of the patients such as age, gender, body mass index and occupation will be recorded. The pain intensity of the patients will be evaluated with the Visual Analog Scale (VAS), their disability with the Oswestry disability index, their kinesiophobia with the Tampo scale for kinesiophobia (TSK), and their quality of life with the SF 36 quality of life scale. TSK is a 17-question scale developed to measure the fear of movement/re-injury. The scale has four answer options rated on a Likert scale (1=Strongly Disagree, 2=Disagree, 3=Agree, 4=Strongly Agree). The total score varies between 17 and 68. Oswestry disability index will be used to measure the person's level of functional disability in individuals with low back pain. Oswestry disability index includes ten subheadings: severity of pain, personal care, lifting loads, walking, sitting, standing, sleeping, sexual life, social life and travel. Each question is given a score between 0 (no disability) and 5 (full disability). The total score varies between 0 (no disability) and 50 (full disability). As the total score increases, functional status worsens. SF-36 short form index will be used to measure quality of life. SF 36 Short form is a questionnaire that provides wide-angle measurement within the quality of life scales and has a generic criterion feature. It consists of 36 questions in 8 categories under the headings of physical function, physical role difficulty, social function, mental health, vitality, pain, emotional role difficulty and general health. The answers to the questions are added as positive and negative and the total score varies between 0 and 100. A high score indicates good health.

ELIGIBILITY:
Inclusion Criteria:

1. Having mechanic lower back pain lasting more than 12 weeks
2. VAS score ≥4
3. Being between the ages of 18-75

Exclusion Criteria:

1. Having inflammatory lower back pain
2. Presence of oncological disease
3. Pregnancy
4. Presence of infection
5. Presence of recent trauma and/or lumbar fracture affecting the lumbar spine
6. Presence of neurological disease that will affect movement
7. Presence of rheumatic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic mechanic low back pain
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia in patients with chronic low back pain | 3 months
  Kinesiophobia will be assessed using the Turkish version of the Tampa Scale for kinesiophobia (TSK). TSK is a 17-question scale developed to measure the fear of movement/re-injury. The scale has four answer options rated on a Likert scale (1=Strongly Disagree, 2=Disagree, 3=Agree, 4=Strongly Agree). The total score varies between 17 and 68.
Disability in patients with chronic low back pain | 3 months
  Oswestry disability index will be used to measure the person's level of functional disability in individuals with low back pain.Oswestry disability index is a test that measures the level of functional disability in individuals with low back pain. It includes ten subheadings: severity of pain, personal care, lifting loads, walking, sitting, standing, sleeping, sexual life, social life and travel. Each question is given a score between 0 (no disability) and 5 (full disability). The total score varies between 0 (no disability) and 50 (full disability). As the total score increases, functional status worsens.
Quality of life in patients with chronic low back pain | 3 months
  SF-36 short form index will be used to measure quality of life. SF 36 Short form is a questionnaire that provides wide-angle measurement within the quality of life scales and has a generic criterion feature. It consists of 36 questions in 8 categories under the headings of physical function, physical role difficulty, social function, mental health, vitality, pain, emotional role difficulty and general health. The answers to the questions are added as positive and negative and the total score varies between 0 and 100. A high score indicates good health.

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Doğan, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Feyza Akan Begoglu, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Gulcan Ozturk, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Meryem Yilmaz Kaysin, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Feyza Unlu Ozkan, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; Ilknur Aktas, Study Chair — Fatih Sultan Mehmet Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No